CLINICAL TRIAL: NCT06001710
Title: Assessment of Needleless Jet Injection in Pain and Anxiety Management During Vital Pulpotomy of Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Jet injector anesthesia
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classic inferior alveolar nerve block anesthesia (Active Comparator): Inferior alveolar nerve block (IANB) is a technique of dental anesthesia, used to produce anesthesia of the mandibular teeth, gingivae of the mandible and lower lip. The conventional IANB is the most commonly used the nerve block technique for achieving local anesthesia for mandibular surgical procedures using long needle
  Interventions: Device: Needleless jet injector
- needleless jet injector anesthesia (Experimental): Jet injection technology uses mechanical energy to force a liquid drug into subcutaneous tissues without a needle using infiltration technique
  Interventions: Device: Needleless jet injector

INTERVENTIONS:
Device: Needleless jet injector — Device consist of injection pen, ampule and activator.

SUMMARY:
To evaluate and compare the efficiency of needleless jet injection versus traditional inferior alveolar nerve block anesthesia in management of pain and anxiety during vital pulpotomy of lower second primary molars using Wong-Baker FACES Pain Rating Scale and Venham's anxiety and behavioral rating scale..

DETAILED DESCRIPTION:
One of the most effective ways to control pain during invasive dental procedures is the use of local anesthesia which considers the most painful phase of treatment. The idea of receiving an injection is fear-inducing for many individuals, both children and adults which can lead patients to avoid dental treatments. Although such fears are outside the control of dentists, some treatment aspects can be modified to increase patient comfort.(1)

Dental care may be associated with pain which may be intertwined with fear and anxiety, especially among children with treatment needs. The pain intensity is multiplied by having higher dental anxiety, a disability, age less than 14 years old and gender (female). The young patient's pain expectations may also add to the situational complexity. Consequently, dental health care may be perceived as insurmountable problem. (2) Administrating an anesthetic agent with a traditional syringe causes discomfort during the puncture and injection stages. (3) Incorrect handling of the syringe is a determining factor for pain (4), which is exacerbated due to excessive pressure on the plunger and rapid injection of large volumes of anesthetic solution.(5)

To minimize the painful sensation during local anesthesia, other methods can be adopted, such as applying topical anesthetics prior to injection (6), using computerized injection systems, and using needleless jet injection systems (7). A needleless system includes a spring coupled to an apparatus that generates sufficient Pressure to (8) push the plunger of the ampoule (9)and makes the anesthetic solution pass through a micro orifice at high speed.

The absence of a needle in a jet injection can result in a more comfortable experience, as this eliminates the puncture and injection phases, which are considered the most painful steps during traditional anesthesia (3). This difference is important as approximately one in five adults have phobia of dental anesthesia due to fear of injections, which leads to interruption of dental treatment (10).

Since there are no studies about the efficacy of needleless jet injection systems during pulpotomy of lower second primary molars, the aim of this clinical trial was to evaluate and compare the efficiency of needleless jet injection versus traditional inferior alveolar nerve block anesthesia in management of pain and anxiety during vital pulpotomy of lower second primary molars

ELIGIBILITY:
Inclusion Criteria:

1. Apparently healthy children.
2. Children aged from 4-8 years old.
3. Both boys and girls were included
4. Children scored (2 or 3) Frankle behavior rating scale.
5. Children had bilateral deep carious lower second primary molars indicated clinically and radiographically for vital pulpotomy
6. Informed consent was included from parents or caregivers.

Exclusion Criteria:

1. Children with evidence of allergy to any materials used in this study
2. Clinical criteria:

   Clinical history of spontaneous pain, intra-oral facial swelling or presence of fistula or sinus tract.

   Tooth with irreversible pulpitis, determined as continuous bleeding exceeding 5 minutes, dark to purple blood color or pulp necrosis.
3. Radiographic criteria:

Presence of any signs of internal or external root resorption, furcation radiolucency or periapical pathosis as revealed by preoperative periapical radiography.

-

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Wong-Baker FACES Pain Rating Scale | After local anesthesia and during pulpotomy
  a method for someone to self-assess and effectively communicate the severity of pain they may be experiencing. The scale contains a series of six faces ranging from a happy face at 0 to indicate "no hurt" to a crying face at 10 to indicate "hurts"
Venham's anxiety and behavioral rating scale | After local anesthesia and during pulpotomy
  assess the anxiety and uncooperative behavior of children in the dental setting.consist of five behavioral defined categories ranging from 0 to 5 with higher score, indicating greater level of anxiety or lack of cooperation.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine , Suez Canal University, Ismailia, Egypt